CLINICAL TRIAL: NCT05138536
Title: Does Comprehensive CT Change Management in Trauma Patients with No Neurologic Deficits
Brief Title: CT Change Management in Trauma Patients
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 024.TRA.2016.D
Record Dates: First submitted 2019-04-03; First posted 2021-12-01 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Trauma; Neurologic Deficits
MeSH Terms: conditions — Wounds and Injuries; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Pan-Computer Tomography — trauma centers use the pan-computed tomography (CT) scan (head, neck, chest, and abdomen/pelvis) for the evaluation of blunt trauma.

SUMMARY:
In high-volume trauma centers, multi-slice CT scanners have become the routine imaging modality for screening trauma patients due to their speed and accuracy. In trauma patients with no known neurologic deficits, diagnostic CT is often obtained though it remains unclear whether this affects management of the patient [1]. With the growing cost of health care, a careful look at the benefit and cost of CT is needed to determine how to best utilize this modality in the evaluation of trauma patients.

HYPOTHESIS: In trauma patients with absence of neurologic defects, the addition of comprehensive CT does not change overall clinical management.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to determine the benefit of the CT scan in the clinical management or outcomes of the trauma patients with no neurologic deficits.

Primary Outcome: Percentage of trauma patients with no known neurologic deficits who underwent a CT, any clinically impactful CT findings.

Secondary Outcome: Percentage of benefits CT provides in clinical features, clinical outcomes, injury severity score, GCS, age, sex, ethnicity, cause of injury, mechanism of injury, hospital length of stay, operative vs. non-operative, discharge disposition, radilogy, pathology results and images, any additional morbidities, total cost, 30-day readmission rate, and morality. And when operation does occur, the types of operation and the resulting cost and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18-years-old
* No localizing neurologic defect
* Any cause or mechanism of injury
* Comprehensive CT obtained

Exclusion Criteria:

• Any patients that are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All trauma patients from Methodist Health System.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of trauma patients with no known neurologic deficits who underwent a CT | April 2006 - April 2016
  the benefit of pan-CT with no neurologic deficits

SECONDARY OUTCOMES:
Percentage of benefits CT provides in clinical features | April 2006 - April 2016
  Clinical outcomes, injury severity score, GCS, age, sex, ethnicity, cause of injury, mechanism of injury, hospital length of stay, operative vs non-operative

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Amos, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided